CLINICAL TRIAL: NCT05861908
Title: Impact of Placement Techniques on Three-year Clinical Performance of Class II Bulk-fill Resin Composite Restorations and Laboratory Investigation of Marginal Adaptation
Brief Title: Bulk-fill With Different Technique Three-year Clinical Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M01060421
Record Dates: First submitted 2023-03-29; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-03

CONDITIONS: Bulk-fill Which is Special Type of Resin Composite; Bisphenol A-Glycidyl Methacrylate

STUDY DESIGN:
Intervention Model Description: Multi-arm parallel design was followed in this study. There were four group according to placement techniques of bulk-fill resin composite restorations. Each group received 20 restored class II cavities.
  All the restorations will be clinically evaluated after 1 week(baseline), 12, 24 and 36 months. Restoration will be evaluated using FDI criteria
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Body Bulk-Fill (Experimental): 20 cavity class II restored with Body bulk-fill Resin composite
  Interventions: Other: Filtek™ Bulk Fill restoration
- preheated Bulk-Fill (Experimental): 20 cavity class II restored with preheated bulk-fill Resin composite
  Interventions: Other: Heated Filtek™ Bulk Fill restoration
- Injectable Bulk-Fill (Experimental): 20 cavity class II restored with injectable bulk-fill Resin composite
  Interventions: Other: G-aenial™ BULK Injectable restoration
- Sonic-Fill (Experimental): 20 cavity class II restored with sonic-fill bulk-fill Resin composite
  Interventions: Other: Sonicfill3 restoration

INTERVENTIONS:
Other: Filtek™ Bulk Fill restoration — restoration of class II caries with different bulk-fill technique
  Arms: Body Bulk-Fill
Other: Heated Filtek™ Bulk Fill restoration — restoration of class II caries with different bulk-fill technique
  Arms: preheated Bulk-Fill
Other: G-aenial™ BULK Injectable restoration — restoration of class II caries with different bulk-fill technique
  Arms: Injectable Bulk-Fill
Other: Sonicfill3 restoration — restoration of class II caries with different bulk-fill technique
  Arms: Sonic-Fill

SUMMARY:
The current study will be intended to evaluate and compare three-year clinical performance of class II bulk-fill resin composite restorations placed with different techniques.

DETAILED DESCRIPTION:
Fifty patients with proximal carious lesion in permanent molars were included in the study. A total eighty class II cavities were restored with one of the following bulk-fill resin composite with their adhesive systems (n=20) Filtek™ Bulk Fill, Heated Filtek™ Bulk Fill, G-aenial™ BULK Injectable or Sonicfill3. Double blinded randomized clinical trial with survival and clinical quality were evaluated at baseline, after 12 , 24 and 36months using modified FDI(Fédération dentaire internationale) World Dental Federation criteria

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Good oral hygienic
* Patient aging 18-35 year
* Patient available for follow-up visits compound class II (mesio-occlusal or disto-occlusal)
* Carious lesion in the external and middle third of dentin thickness
* ICDAS (International caries detection and assessment system) 4 or 5 that diagnosed clinically and radiographically.
* Maxillary or mandibular first or second molars
* Tooth with antagonist and adjacent mesial and distal tooth contact,
* Normal response to a vitality test.

Exclusion Criteria:

* Poor oral hygiene
* Severe or chronic periodontitis
* Heavy bruxism
* Occlusion fewer than 20 teeth
* Sensitivity to resin-based material.
* Patients with orthodontic treatment
* Patients on pregnancy or lactation
* chronic use of anti-inflammatory drugs, analgesic, and/or psychotropic drugs
* Patient potentially unable to attend recall visits
* Teeth would need direct pulp capping or
* Teeth act as abutment for fixed or removable prosthesis.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-05-09 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2024-05-09 (Estimated)

PRIMARY OUTCOMES:
Esthetic Properties of restorations | Three years Follow up
  criteria that evaluated according to Modified FDI(International Dental Federation) world dental federation is:
  1. Surface luster
  2. Staining
  3. Color match and translucency
  4. Esthetic and Anatomic form
  Descriptive scale from 1 to 5. Note: 1 is clinically excellent 5 is clinically poor
Functional Properties of restorations | Three years Follow up
  criteria that evaluated according to Modified FDI (International Dental Federation) world dental federation is:
  1. Fractures of material and retention
  2. Marginal adaptation
  3. Occlusal contour and wear
  4. Proximal anatomical form
  5. Patient's view
  Descriptive scale from 1 to 5. Note: 1 is clinically excellent 5 is clinically poor
Biological Properties of restorations | Three years Follow up
  criteria that evaluated according to Modified FDI (International Dental Federation) world dental federation is:
  1. Post-operative (hyper-sensitivity) and tooth vitality
  2. Recurrence of caries, erosion, abfraction
  3. Tooth integrity (enamel cracks, tooth fractures)
  4. Periodontal
  5. Adjacent Mucosa
  6. Oral and General Health
  Descriptive scale from 1 to 5. Note: 1 is clinically excellent 5 is clinically poor

CONTACTS AND LOCATIONS:
Locations (1):
- Operative Department, Faculty of Dentistry, Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided